CLINICAL TRIAL: NCT06223204
Title: GLEAM: Noninvasive Glucose Measurement Using Impedance Tomography - a Pilot Project
Brief Title: GLEAM: Noninvasive Glucose Measurement Using Impedance Tomography
Acronym: GLEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: CSEM Centre Suisse d'Electronique et de Microtechnique SA (Unknown); Idiap Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GLEAM
Record Dates: First submitted 2023-12-19; First posted 2024-01-25 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled euglycemia, hypoglycemia and hyperglycemia (Other)
  Interventions: Other: Controlled euglycemia, hypoglycemia and hyperglycemia

INTERVENTIONS:
Other: Controlled euglycemia, hypoglycemia and hyperglycemia — EIT measurements are collected in different glycemic states (euglycemia, hypoglycemia and hyperglycemia). Venous blood glucose is measured using a gold-standard glucose analyzer.

SUMMARY:
The GLEAM study aims at assessing the potential of electrical impedance tomography (EIT) for noninvasive glucose measurement.

DETAILED DESCRIPTION:
Within the GLEAM study, paired samples of EIT and blood glucose measurements will be collected in individuals with type 1 diabetes during standardized euglycemia, hypoglycemia and hyperglycemia. These samples will be used to assess the potential of EIT for noninvasive glucose measurement and/or dysglycemia detection.

ELIGIBILITY:
Inclusion Criteria:

* Written, informed consent
* Type 1 Diabetes mellitus as defined by WHO for at least 6 months
* Aged 18 - 60 years
* HbA1c ≤ 9.0 %
* Insulin treatment with good knowledge of insulin self-management
* Use of a continuous (CGM) or flash glucose monitoring system (FGM)
* Native language German or Swiss German

Exclusion Criteria:

* Incapacity to give informed consent
* Contraindications to insulin aspart (NovoRapid®)
* Known allergies to adhesives of the EIT device (e.g., gel electrodes)
* Pregnancy, breast-feeding or lack of safe contraception
* Active heart, lung, liver, gastrointestinal, renal or psychiatric disease
* Patients with implantable electronic devices (e.g., pacemaker or implantable cardioverter defibrillator (ICD)) or thoracic metal implants
* Epilepsy or history of seizure
* Active drug or alcohol abuse
* Chronic neurological or ear-nose-and-throat (ENT) disease influencing voice or history of voice disorder
* Thoracic or back deformities
* Body mass index (BMI) >35.0 kg/m2
* Open wounds, burns, or rashes on the upper thorax
* Active smoking
* Medication known to interfere with voice or to induce listlessness (e.g., opioids, benzodiazepines, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Change of the electrical impedance tomography (EIT) signal of the thoracic region across the glycemic trajectory. | 5 hours
  EIT signals will be collected at multiple frequencies between 50 kHz and 1 MHz from the thoracic region in euglycemia, hypoglycemia and hyperglycemia using a multi-channel EIT measurement device.

SECONDARY OUTCOMES:
Change of hypoglycemia symptoms across the glycemic trajectory. | 5 hours
  Hypoglycemia symptoms will be collected in euglycemia, hypoglycemia and hyperglycemia using a standardized questionnaire (Edinburgh Hypoglycemia Scale, a higher score means more symptoms, minimum score 7 points, maximum score 77 points).
Voice parameters indicative of dysglycemia | 5 hours
  Voice data will be collected using a microphone in euglycemia, hypoglycemia and hyperglycemia. After sampling, an interpretable machine learning (ML) method will be used to identify voice parameters indicative of dysglycemia.
Change in cognitive performance across the glycemic trajectory. | 5 hours
  Cognitive performance will be assessed using the Trail Making B Test (more time needed to complete the tests means worse cognitive performance).
Change in cognitive performance across the glycemic trajectory. | 5 hours
  Cognitive performance will be assessed using the Digit Symbol Substitution Test (higher score means better cognitive performance).
Performance of a machine learning model to detect dysglycemia from the above-mentioned signals (EIT, symptoms, voice, physiological signals) quantified as area under the receiver operating characteristics curve (AUROC). | 5 hours
  Signals for machine learning modeling will be collected in euglycemia, hypoglycemia and hyperglycemia.
Performance of a machine learning model to detect dysglycemia from the above-mentioned signals (EIT, symptoms, voice, physiological signals) quantified as sensitivity. | 5 hours
  Signals for machine learning modeling will be collected in euglycemia, hypoglycemia and hyperglycemia.
Performance of a machine learning model to detect dysglycemia from the above-mentioned signals (EIT, symptoms, voice, physiological signals) quantified as specificity. | 5 hours
  Signals for machine learning modeling will be collected in euglycemia, hypoglycemia and hyperglycemia.
Performance of the machine learning model to predict glucose values from the above-mentioned signals (EIT, symptoms, voice, physiological signals) quantified as root mean squared error (RMSE). | 5 hours
  Signals for machine learning modeling will be collected in euglycemia, hypoglycemia and hyperglycemia.
Performance of the machine learning model to predict glucose values from the above-mentioned signals (EIT, symptoms, voice, physiological signals) quantified as mean absolute relative difference (MARD). | 5 hours
  Signals for machine learning modeling will be collected in euglycemia, hypoglycemia and hyperglycemia.
Performance of the machine learning model to predict glucose values from the above-mentioned signals (EIT, symptoms, voice, physiological signals) using Bland-Altman plots. | 5 hours
  Signals for machine learning modeling will be collected in euglycemia, hypoglycemia and hyperglycemia.
Performance of the machine learning model to predict glucose values from the above-mentioned signals (EIT, symptoms, voice, physiological signals) using the Clarke Error Grid. | 5 hours
  Signals for machine learning modeling will be collected in euglycemia, hypoglycemia and hyperglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, Prof. MD, Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism; Bern, Switzerland
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No